CLINICAL TRIAL: NCT00495105
Title: Dairy Foods and Blood Pressure in Multi-Ethnic Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Debra K. Sullivan, PhD, RD (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor-Investigator, Debra K. Sullivan, PhD, RD, Chair, Midwest Dairy Professor of Clinical Nutrition, University of Kansas Medical Center
Organization: University of Kansas Medical Center (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 1R01HL080967-01A2 (NIH); 8586; 1R01HL080967-01A2 (NIH)
Record Dates: First submitted 2007-06-27; First posted 2007-07-02 (Estimated); Last update posted 2013-02-12 (Estimated); Status verified 2013-02

CONDITIONS: Blood Pressure, High
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Two Servings of Dairy Snacks (Experimental): Intervention group received two servings of dairy food per day as a snack at school for 6 months as well as nutrition education.
  Interventions: Behavioral: Two Servings of Dairy Snacks
- No Dairy Snacks (No Intervention): Control Group did not receive any snacks or education.

INTERVENTIONS:
Behavioral: Two Servings of Dairy Snacks — 2 servings of dairy products as snacks at school to third, fourth, and fifth grade students each day for 24 weeks. The serving size of each dairy snack is based on its calcium content with the goal of adding an extra 300 mg of calcium to the intervention group's daily intake.
  Arms: Two Servings of Dairy Snacks

SUMMARY:
To prevent excess increases in blood pressure in children by providing two servings of dairy foods as snacks daily at school. We hypothesize that children who receive the two dairy snacks will exhibit significantly less of an increase in blood pressure over six months as compared to control children.

DETAILED DESCRIPTION:
The primary aim of the study is to determine the impact of dairy foods on blood pressure; however, we will also evaluate the effect of the intervention on body weight and composition. Specifically, we will evaluate change in body mass index (BMI, kg/m2], waist circumference in all subjects and body composition by bioelectrical impedance (BIA) in a subset. We hypothesize that children receiving the dairy snacks will exhibit less increase in BMI and body fat than control subjects. We are studying a group of children at high risk for elevated blood lipids and glucose intolerance due to their racial/ethnic makeup and high prevalence of overweight and obesity. Thus, we will evaluate the impact of the intervention on blood lipids, glucose and insulin in a subset of subjects.

We hypothesize that children receiving the dairy foods will exhibit improvements in their lipids, glucose and insulin as compared to control children. We also plan to determine their eating habits through a 24 hour dietary recall at the beginning, middle and end of the study, with 2 additional recalls for the subset at each time point. Dietary behavior and self efficacy will be analyzed before and after the intervention through a questionnaire. Physical activity levels will be assessed by a short physical activity questionnaire on all students and through the utilization of accelerometers in the subset. Our control schools will undergo the same testing, but will not receive any intervention.

ELIGIBILITY:
Inclusion Criteria:

* Willingness to participate in the study
* Signed informed consent form by the parents and/or guardians
* Assent from the child

Exclusion Criteria:

* Children with food allergies or other dietary requirements that restrict their ability to consume the snack
* Children with a chronic medical condition that may influence blood pressure or calcium metabolism such as renal disease or type 1 diabetes mellitus

Ages: 8 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 2115 (Actual)
Dates: Start 2007-08; Primary Completion 2009-05 (Actual); Study Completion 2009-05 (Actual)

PRIMARY OUTCOMES:
Blood Pressure Measurements | 0, 3 and 6 Months

SECONDARY OUTCOMES:
Body Composition Measurements | 0, 3 and 6 Months
Dietary intake | 0, 3 and 6 Months
Blood Glucose, insulin, lipid profiles, and physical activity measurements by questionnaire and accelerometers to 10% of study population | 0 and 6 Months

CONTACTS AND LOCATIONS:
Overall Officials: Debra K. Sullivan, PhD, RD, LD, Principal Investigator — University of Kansas Medical Center
Locations (1):
- University of Kansas Medical Center, Kansas City, Kansas, United States